CLINICAL TRIAL: NCT02509169
Title: Trans-catheter Arterial p53-gene-embolization Using Gelatin Sponge Particles in Treatment of Patients With Advanced Hepatocellular Carcinoma: A Phase II Study
Brief Title: Trans-catheter Arterial Embolization Combined With p53 Gene Therapy for Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAp53-110
Record Dates: First submitted 2015-07-19; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Genes, p53

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAE plus p53 gene (Experimental): Trans-catheter embolization (TAE) combined with recombinant adenoviral human p53 gene (rAd-p53) will be given one per month
  Interventions: Drug: TAE plus P53 gene
- TAE (Active Comparator): Trans-catheter embolization (TAE) will be given once per month
  Interventions: Other: TAE

INTERVENTIONS:
Drug: TAE plus P53 gene — Trans-catheter embolization combined with recombinant adenoviral human p53 gene therapy
  Arms: TAE plus p53 gene
Other: TAE — Trans-catheter embolization
  Arms: TAE

SUMMARY:
An open-labeled, randomized, active-controlled phase II study to investigate clinical efficacy and immunoreaction using trans-catheter arterial embolization (TAE) combined with p53 gene therapy in treatment of advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Treatment options for advanced HCC are limited due to patients' poor condition, advanced stage, concomitant intra- and extra-liver diseases, and resistance to both chemo- and radio-therapy. Trans-catheter embolization (TAE) is a safe locoregional treatment for advanced HCC and p53 gene has multiple anticancer functions, and both methods do not have immune-inhibitory effects as chemo- or radio-therapy. The objectives of this study are to investigate clinical efficacy and immunoreaction usingTAE plus recombinant adenoviral human p53 gene (rAd-p53) in treatment of advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically diagnosed unresectable HCC
* over 18 years old
* with an Eastern Cooperative Oncology Group (ECOG) score of 0-2
* with Barcelona Clinic Liver Cancer (BCLC) Stage of B or C
* with Child-Pugh score A or B; with normal tests of hemogram, blood coagulation, liver and kidney function
* signed the informed consent form.

Exclusion Criteria:

* hypersensitive to study drug
* With an abnormal coagulation condition or bleeding disorder
* infections
* with serious conditions which prevent using the study treatment
* pregnant or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years
  overall survival will be follow up to 2 years

SECONDARY OUTCOMES:
immuno-reaction (lymphocyte counts and subgroup ratios) | 3 months
  The immune reaction after study treatment will be assessed every one week until 3 months after the first treatment
progression free survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- first affiliated hospital in Dalian University, Dalian, Liaoning, China